CLINICAL TRIAL: NCT07079345
Title: PET/MR Multimodal Quantitative Imaging of Cerebral Ischemia With CBF and CMRGlc Assessment in Cephalo-Carotid Atherosclerosis
Brief Title: PET/MR Multimodal Quantitative Analysis of CBF and CMRGlc in Cerebral Ischemia
Acronym: PMQIC
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: LYS[2025]201-001; 2024ZD0539800 (Other Grant/Funding Number: Noncommunicable Chronic Diseases-National Science and Technology Major Project)
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: PET/MR; Stroke Ischemic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
Research Purpose:

This project focuses on clinical research issues in the diagnosis, treatment, and evaluation of patients with cephalic and carotid atherosclerosis. Through multimodal imaging technology, it aims to optimize non-invasive quantitative algorithm models for cerebral blood flow and cerebral metabolism, explore new imaging markers, and investigate quantitative indicators of cerebral blood flow and metabolism for the diagnosis, treatment, and evaluation of patients with cephalic and carotid atherosclerosis undergoing drug therapy or surgical treatment.

Research Design:

1. Study Type: Observational study
2. Study Subjects: In accordance with the *Chinese Clinical Management Guidelines for Cerebrovascular Diseases (2nd Edition)*, patients with cephalic and carotid atherosclerotic stenosis admitted to the department of neurosurgery will be enrolled. Data collection time points are at enrollment, 6-month follow-up, and 12-month follow-up.
3. Sample Size: 200 patients with cephalic and carotid atherosclerotic stenosis.
4. Observation Indicators: Distribution patterns of cerebral blood flow and metabolic reduction areas in patients; correlation analysis between blood flow, metabolic values and clinical scores.
5. Statistical Analysis Methods: Statistical analysis will be performed using Statistical Package for the Social Sciences (SPSS) version 21.0. All statistical results will be expressed as mean ± standard deviation. First, the Shapiro-Wilk test will be used to assess normal distribution. Under the premise of normal distribution, paired t-test will be used to compare blood flow and metabolic values between the lesion area and the contralateral area of patients, as well as to compare changes in blood flow and metabolism of patients at different time points. Pearson correlation analysis will be used to analyze the relationship between blood flow/metabolic parameters and clinical neurological function scores. The Mann-Whitney U test will be used to analyze variables with non-normal distribution. A P value < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Angiography diagnosed unilateral anterior circulation head carotid artery stenosis, the diameter of the tube was reduced by >70%, and the contralateral anterior circulation and bilateral posterior circulation did not exceed the stenosis of >50% of the diameter reduction;
2. Must have had a transient ischemic attack or ischemic stroke within the area of the diseased vessel within the past 12 months, with the most recent onset being more than 3 weeks;
3. MRI showed no new infarct lesions in the skull;
4. There is no infarct lesion in the previous pontine area;
5. Research participants and informants can complete relevant examinations and follow-ups;
6. Informed consent signed by the study participant or his/her authorized representative;

Exclusion Criteria:

1. Poor image quality caused by head movement or other reasons during scanning
2. Presence of other neurological diseases that can cause brain dysfunction (such as depression, brain tumor, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal pressure hydrocephalus, etc.)
3. Presence of other systemic diseases that can cause cognitive impairment, such as hepatic insufficiency, renal insufficiency, thyroid dysfunction, severe anemia, folic acid and vitamin B12 deficiency, specific infections (such as syphilis, HIV), alcohol and drug abuse, etc
4. Presence of other known diseases that may cause cognitive impairmentPresence of other known diseases that may cause cognitive impairment
5. Individuals with severe visual or hearing impairment, claustrophobia, or other conditions that prevent cooperation with MRI examination
6. Individuals suffering from diseases that make it impossible to cooperate with cognitive examinations
7. Refusal to sign the informed consent form at baseline

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with intracranial artery stenosis due to head and carotid atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the cerebral blood flow (CBF, mL 100g-1 min-1) at 6 Months | CBF and CMRGlc at 6 months post-treatment
  Results of integrated PET/MR examination at 6 months post-treatment
Change from Baseline in the cerebral metabolic rate of glucose (CMRglc, μmol 100g-1 min-1) at 6 Months | CBF and CMRGlc at 6 months post-treatment
  Results of integrated PET/MR examination at 6 months post-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospitail, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No